CLINICAL TRIAL: NCT01839669
Title: The CurePPaC Study - Analysing Non-surgical Treatment Strategies to Cure Pes Planovalgus Associated Complaints
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Not possible to enroll enough patients in reasonable time.
Sponsor: Bern University of Applied Sciences (Other)
Collaborators: Swiss National Science Foundation (Other); Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Principal Investigator, Heiner Baur (PhD), PhD, Bern University of Applied Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 140928
Record Dates: First submitted 2013-04-17; First posted 2013-04-25 (Estimated); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Foot Injuries; Posterior Tibial Tendon Dysfunction
Keywords: conservative therapy; Foot-Function-Index; functional movement changes; non-surgical treatment; pes planovalgus; posterior tibial tendon dysfunction
MeSH Terms: conditions — Foot Injuries; Posterior Tibial Tendon Dysfunction; Clubfoot | interventions — Foot Orthoses

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Foot Orthoses Only (Active Comparator): including Patient Education; Abbreviation: FOO
  Interventions: Device: Foot Orthoses Only
- Foot Orthoses and Eccentric Exercise (Experimental): including Patient Education; Abbreviation: FOE
  Interventions: Procedure: Foot Orthoses and Eccentric Exercise
- Sham Foot Orthoses (Sham Comparator): including Patient Education; Abbreviation: FOS
  Interventions: Device: Sham Foot Orthoses

INTERVENTIONS:
Device: Foot Orthoses Only — patients wear foot orthoses as a treatment condition - no further therapy
  Arms: Foot Orthoses Only
Procedure: Foot Orthoses and Eccentric Exercise — patients wear foot orthoses and they perform an additional home-based eccentric training program for the M. tibialis posterior
  Arms: Foot Orthoses and Eccentric Exercise
Device: Sham Foot Orthoses — patient wear sham foot orthoses (control condition)
  Arms: Sham Foot Orthoses

SUMMARY:
Pes planovalgus, also called flat foot, is a common foot deformity characterized by a flattening of the foot's longitudinal arch and is accompanied by a dysfunction of the posterior tibial tendon ("posterior tibial tendon dysfunction" or "PTTD"). Early stages of this pathology are thought to be treated with non-surgical therapy options like foot orthoses (relief of tendon stress by mechanical unloading of the arch), strengthening exercises or basic physiotherapeutic measures. Recent literature clearly states the urgent need for high quality studies to evaluate the proposed non-surgical treatments (Bowring 2009, 2010). There is only one high quality study available that shows benefits of orthoses therapy and exercise (Kulig 2009). No study to date evaluated functional changes pre-post in dynamic movement pattern like gait or stair climbing. The widespread use of several non-surgical treatment strategies lead to extensive financial expenses of the health care system. An optimized therapeutic strategy could eventually lead to more efficient health care investments. The presented proposal addresses this latest knowledge and aims to analyse non-surgical treatment strategies to Cure Pes Planovalgus associated Complaints (CurePPaC) in the CurePPaC Study.

DETAILED DESCRIPTION:
Introduction: Pes planovalgus or flatfoot-associated complaints are frequent symptoms, which are thought to be caused by the foot deformity itself. Concurrently, the multifactorial weakness of the M. tibialis posterior and its tendon (trauma, systemic disease, chronic tendon degeneration by overuse) can lead to a flattening of the medial longitudinal arch of the foot. Affected patients suffer from functional impairment and pain. Less severe cases are eligible for non-surgical treatment. Foot orthoses are considered to be the first line approach. Furthermore strengthening of the arch and ankle stabilizing muscles are thought to contribute to an active compensation of the deformity. There is only limited evidence concerning the numerous therapy approaches since high quality studies are missing. One excellent report (Kulig et al. 2009) shows clear benefits by the use of foot orthoses and eccentric strengthening exercises. Beside the fact that evidence-based guidelines for therapy have yet to be developed, no data is available showing functional benefits that accompany the therapy process. This would give further insight into mechanisms behind non-surgical management strategies and how patients benefit functionally from therapy. Purpose: The purpose of this randomized longitudinal intervention study is the evaluation of the therapeutic benefit of three different non-surgical treatment regimens (foot orthoses only FOO, foot orthoses and eccentric exercise FOE, foot orthoses sham treatment FOS) in patients with Pes planovalgus and accompanying complaints. Furthermore the analysis of possible functional changes in gait mechanics (kinematic and kinetic view) and neuromuscular control (electromyographic analysis) will contribute to a superior understanding of functional changes that accompany non-operative management. The purpose of the study is to optimize non-surgical management in patients suffering from Pes planovalgus associated pain leading to an efficient use of health care system's financial resources. Methods: 60 patients with Pes planovalgus associated complaints (clinical diagnosis with plain weight bearing radiographs), M. tibialis posterior dysfunction) are included in the study. Functional impairment is evaluated pre and post intervention by the Foot-Function-Index (FFI, German version). Anthropometric data recording is followed by preparation of subject's foot anatomical landmarks with retroreflective markers and superficially detectable muscles of the ankle joint complex are prepared with surface electromyography (SEMG) electrodes. The 3D kinematic data allows inter alia the calculation of segmental angels of the lower extremity and measurement of navicular drop. The neuromuscular activity is analysed in the time (on-off pattern) and amplitude domain (gait cycle specific phases). Procedure: Potential participants are recruited via the Outpatient Clinic of the Department of Orthopaedic Surgery of the Inselspital, University Hospital, Bern. After initial screening, subjects are randomized to one of three intervention groups (foot orthoses only FOO, foot orthoses and eccentric exercise FOE, foot orthoses sham treatment FOS). FOO-subjects wear custom-made foot orthoses only. FOE-subjects wear individually accustomed foot orthoses and they will perform a combined monitored and home training program to progressively strengthen the M. tibialis posterior and accompanying ankle stabilizing muscles with eccentric exercises. FOS-subjects wear custom-made sham foot orthoses without the functional elements of the treatment orthoses (longitudinal arch support, ankle stabilizer, bowl-shaped heel for rearfoot stability). Subjects are measured pre and post intervention (12 weeks). Measurements include the primary outcome measure Foot-Function-Index (FFI, German version: total score) followed by basic anthropometric measures. Subject preparation allows then the measurement of 10 trials on a walkway and on stairs with embedded force plates in barefoot condition. An average step cycle out of 10 trials is calculated and biomechanical outcome measures are extracted. A re-test allows the calculation of intervention effects by one-factor ANOVA (group: treatment FOO vs. FOE vs. FOS) for repeated measures.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-60
* Current complaint of foot and ankle pain that lasted for 3 months or more
* Flexible Pes planovalgus deformity in the clinical assessment
* Posterior tibial tendon dysfunction (PTTD) of stage I and II (Johnson & Strom 1989)
* Pes planovalgus foot deformity with longitudinal arch flattening verified by radiograph (Younger 2005): Lateral view: lateral talo-first metatarsal angle ≠ 0° (break of axis): angle >10° according to Younger (2005); 60Anteroposterior view: anteroposterior talo-first metatarsal angle ≠ 0° (break of axis): angle >10° according to Younger (2005)
* "too-many toes"-sign from rear frontal view with an abducted forefoot (Johnson & Strom 1989, Kulig 2009b)
* Eligibility for non-surgical treatment
* No indication / not yet an indication for surgical treatment of foot deformity

Exclusion Criteria:

* Rigid foot deformity
* Posterior tibial tendon dysfunction (PTTD) of stage III and IV according to Johnson & Strom 1989 (=>rigid foot deformity)
* Cardio-, neuro-, or peripheral vascular pathology, musculoskeletal pathology, acute infection or alcohol addiction limiting participation in study protocol
* Acute use of local or systemic analgesics
* Acute physical therapy, training therapy or physiotherapy
* Acute overuse or traumatic injury to the lower leg (excluding Pes planovalgus associated pathology)
* Prior surgery to the lower limb

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2013-07; Primary Completion 2017-10-25 (Actual); Study Completion 2017-10-25 (Actual)

PRIMARY OUTCOMES:
Foot Function Index - total score | change from baseline (pre intervention) to week 12 (post intervention)
  additional analysis of change from baseline to week 4, and analysis of change from baseline to week 8

SECONDARY OUTCOMES:
Foot Function Index - subcategory pain | change from baseline (pre intervention) to week 12 (post intervention)
  additional analysis of change from baseline to week 4, and analysis of change from baseline to week 8
Foot Function Index - subcategory disability | change from baseline (pre intervention) to week 12 (post intervention)
  additional analysis of change from baseline to week 4, and analysis of change from baseline to week 8
Foot Function Index - subcategory activity limitation | change from baseline (pre intervention) to week 12 (post intervention)
  additional analysis of change from baseline to week 4, and analysis of change from baseline to week 8

OTHER OUTCOMES:
Pain Disability Index | change from baseline (pre intervention) to week 12 (post intervention)
  additional analysis of change from baseline to week 4, and analysis of change from baseline to week 8
Visual Analogue Scale | change from baseline (pre intervention) to week 12 (post intervention)
  assessing pain pre- and post biomechanical testing / change from baseline to week 12
kinematic data from 3d movement analysis | change from baseline (pre intervention) to week 12 (post intervention)
  regarding distance: navicular drop; regarding angular data (angle at initial contact, max. manifestation during stance, range): foot progression angle, forefoot to rearfoot dorsiflexion, forefoot to rearfoot adduction, forefoot to rearfoot supination, ankle dorsiflexion, ankle adduction, ankle eversion, knee flexion, knee adduction, knee internal rotation, hip flexion, hip adduction, hip internal rotation
neuromuscular activity | change from baseline (pre intervention) to week 12 (post intervention)
  EMG of M. tibialis anterior, M. peroneus longus, M. gastrocnemius lateralis/medialis, M. soleus: onset of activation, time of maximum activation, total time of activation, normalized amplitude in preactivation, normalized amplitude in weight acceptance, normalized amplitude in mid-stance, normalized amplitude in push-off

CONTACTS AND LOCATIONS:
Overall Officials: Heiner Baur, PhD, Principal Investigator — Bern University of Applied Sciences, Switzerland; Heiner Baur, PhD, Principal Investigator — Bern University of Applied Sciences, Health, aR&D Physiotherapy
Locations (6):
- Switzerland (6):
  - Spital Netz Bern Ziegler, Bern
  - Klinik Sonnenhof Bern, Bern
  - Inselspital, University Hospital Bern, Bern
  - Salem Spital Bern, Bern
  - Salem-Spital Orthopädische Klinik Bern, Bern
  - spital STS AG, Thun

REFERENCES:
- [Background] Younger AS, Sawatzky B, Dryden P. Radiographic assessment of adult flatfoot. Foot Ankle Int. 2005 Oct;26(10):820-5. doi: 10.1177/107110070502601006. PMID 16221454
- [Background] Johnson KA, Strom DE. Tibialis posterior tendon dysfunction. Clin Orthop Relat Res. 1989 Feb;(239):196-206. PMID 2912622
- [Background] Kulig K, Reischl SF, Pomrantz AB, Burnfield JM, Mais-Requejo S, Thordarson DB, Smith RW. Nonsurgical management of posterior tibial tendon dysfunction with orthoses and resistive exercise: a randomized controlled trial. Phys Ther. 2009 Jan;89(1):26-37. doi: 10.2522/ptj.20070242. Epub 2008 Nov 20. PMID 19022863
- [Background] Bowring B, Chockalingam N. Conservative treatment of tibialis posterior tendon dysfunction--a review. Foot (Edinb). 2010 Mar;20(1):18-26. doi: 10.1016/j.foot.2009.11.001. Epub 2009 Dec 24. PMID 20434675
- [Background] Bowring B, Chockalingam N. A clinical guideline for the conservative management of tibialis posterior tendon dysfunction. Foot (Edinb). 2009 Dec;19(4):211-7. doi: 10.1016/j.foot.2009.08.001. Epub 2009 Sep 18. PMID 20307479
- [Background] Blasimann A, Eichelberger P, Brulhart Y, El-Masri I, Fluckiger G, Frauchiger L, Huber M, Weber M, Krause FG, Baur H. Non-surgical treatment of pain associated with posterior tibial tendon dysfunction: study protocol for a randomised clinical trial. J Foot Ankle Res. 2015 Aug 14;8:37. doi: 10.1186/s13047-015-0095-4. eCollection 2015. PMID 26279682
- See also: project description in the database of the Swiss National Science Foundation — http://p3.snf.ch/project-140928